CLINICAL TRIAL: NCT00796926
Title: Randomised Controlled Trial to Compare the Efficacy of Systane Ultra and Refresh Drop in the Treatment of Dry Eye in Asian Eyes
Brief Title: Trial to Compare the Efficacy of Systane Ultra and Refresh Drop in the Treatment of Dry Eye in Asian Eyes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Louis Tong (Other Government)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Louis Tong, Clinician-Scientist, Consultant, Singapore National Eye Centre
Organization: Singapore National Eye Centre (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R632/53/2008
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Xerophthalmia; Blepharitis
MeSH Terms: conditions — Xerophthalmia; Blepharitis | interventions — methylacetylene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Experimental): Used four times a day topically to each eye
  Interventions: Drug: Systane Ultra eyedrops
- Refresh (Active Comparator): Used four times a day topically to each eye
  Interventions: Drug: Refresh eye drops

INTERVENTIONS:
Drug: Systane Ultra eyedrops — Four times a day
  Other Names: Systane Ultra, Alcon
  Arms: Systane Ultra
Drug: Refresh eye drops — Four times a day
  Other Names: Refresh, Allergan
  Arms: Refresh

SUMMARY:
Systane Ultra is at least as efficacious and safe as Refresh Tears in Asian people with Dry Eyes

DETAILED DESCRIPTION:
Comparison of efficacy of Systane Ultra and Refresh Tears

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is between 40 and 65 years old.
2. Corneal fluorescein staining present in at least one/five sectors of at least one cornea
3. At least one question out of 6 questions on dry eye symptom present often or all the time.

   based on the Salisbury Eye study by Oliver Schein et al. (Does your eye feel dry, gritty, red, watery, crusted, stuck in the morning?) Please see appendix 1.
4. At least one of the following: TBUT <= 5 s or Schirmer I less than 8 mm in at least one eye
5. Yamaguchi score 2 in at least one sector of one of 4 lids (slight advancement of Marx's line in line with Meibomian orifice)
6. Not using non-lubricant ophthalmic drops within the last 30 days and able to abstain from non-trial topical eye medications for 6 weeks.
7. Use of lubricants during the week before recruitment (ranging from 3 times in the week to less than 6 times a day every day).
8. Able to use saline eyedrops during the 7 day 'washout' evaluative phase, between 3 times over week to less than 6 times a day in all days.

Exclusion Criteria:

1. Known history of thyroid disorders (diagnosed by physician).
2. Known history of Sjogren syndrome or rheumatoid arthritis (diagnosed by physician).
3. No ocular surgery within 6 months and LASIK within 1 year.
4. Any intake of central nervous system and hormonal drugs within last 30 days and inability to withhold such drugs for at least 6 weeks.
5. Ocular surface diseases such as pterygium, or obvious lid/orbital disease with lagophthalmos.
6. Anticipated necessity to wear contact lens in the duration of the study.
7. Not living in the same household as another participant of the study.
8. Any other specified reason as determined by clinical investigator.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, FRCS, MD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Center, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Systane Ultra: four times a day for six weeks in each eye
- Refresh: Four times a day for 6 weeks in each eye
Period: Overall Study
Arm/Group | Systane Ultra | Refresh
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Ultra | Refresh | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (5.8) | 55.7 (5.5) | 55.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Singapore | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Score (VAS)
Description: Global score calculated from square root( square of (discomfort severityX Sqr(symptom frequency)) Scale from 0 to 100 higher value indicates more adverse symptoms each subscale severity or frequency also has same minimum and maximum
Time Frame: 6 weeks
Population: intention to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Systane Ultra | Refresh
Number analyzed (Participants) | 14 | 15
scores on a scale | 21.55 (16.8) | 27.27 (15.0)
Statistical Analysis 1: Comparison: Systane Ultra vs Refresh; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Corneal Fluorescein Staining Score
Description: This is graded in the 5 zones of each cornea according to number of spots of corneal fluorescein staining, confluency of spots and presence of filaments if any
Time Frame: 6 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: staining grade

3. Secondary Outcome: Tear Break Up Time (TBUT)
Time Frame: 6 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: seconds

4. Secondary Outcome: Schirmer I Reading
Time Frame: 6 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mm

5. Secondary Outcome: Meibography Grading
Time Frame: 6 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: arbitrary grade

6. Secondary Outcome: Tear Osmolarity
Description: This is measured by the TearLab (Ocusense) system
Time Frame: 6 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mOsM

7. Secondary Outcome: Superior and Inferior Tear Meniscus Height
Description: This is determined by anterior segment OCT visante system
Time Frame: 6 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mm

ADVERSE EVENTS:
Arm/Group | Systane Ultra | Refresh
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No